CLINICAL TRIAL: NCT00451815
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose Escalation Study of Multiple Oral Dose Administration of BIIB014 in Subjects With Early Parkinson's Disease
Brief Title: BIIB014 Phase 2a Monotherapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 204-PD-201
Record Dates: First submitted 2006-01-31; First posted 2007-03-26 (Estimated); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — 3-(4-amino-3-methylbenzyl)-7-(2-furyl)-3H-(1,2,3)triazolo(4,5-d)pyrimidine-5-amine; Dihydrotachysterol

STUDY DESIGN:
Masking Description: Double

INTERVENTIONS:
Drug: active drug (BIIB014) at 10, 30, 100, or 300 mg once daily.
Drug: placebo

SUMMARY:
To assess the preliminary safety and tolerability of multiple oral doses of BIIB014 in subjects with early PD.

ELIGIBILITY:
Inclusion Criteria:

Unless otherwise specified, to be eligible to participate in this study, candidates must meet the following eligibility criteria at the time of the Baseline Visit (Day -1):

1. Must give written informed consent. Must also provide all authorizations required by local law.
2. Aged 30 to 78 years old at the time of informed consent.
3. If female, must be postmenopausal for at least 1 year, surgically sterile, or willing to practice effective contraception during the study. Nursing mothers, pregnant women, and women planning to become pregnant while on study are to be excluded.
4. Carry a diagnosis of probable idiopathic PD, made by a Movement Disorder Specialist, with asymmetric onset and at least 2 of the following cardinal features of PD: bradykinesia, rigidity, or a classic PD resting tremor.
5. Be Hoehn & Yahr Stage I-III inclusive when OFF.
6. Have a Total Unified PD Rating Scale (UPDRS) OFF score of ³ 8.
7. Have taken no prescribed medications for PD for a minimum of 2 weeks before the Baseline Visit (Day -1).
8. Are willing to abstain from alcohol for the duration of the study.
9. Have no clinically significant baseline ECG (12-lead) and laboratory abnormalities (as determined by the Investigator), unless exempted by the Biogen Idec Medical Director.
10. Agree to provide blood samples for mRNA and DNA analysis, which will be collected and banked and may be used for exploratory pharmacogenomic studies.

Exclusion Criteria

Unless otherwise specified, candidates will be excluded from study entry if any of the following exclusion criteria exist at the time of the Baseline Visit (Day -1):

1. Mini Mental State Examination (MMSE) score <27.
2. History or clinical features such as impaired downward gaze, prominent axial rigidity, gait initiation failure, autonomic dysfunction, etc. consistent with an atypical parkinsonism syndrome.
3. Any significant non-PD central nervous system disorder.
4. Significant AXIS I psychiatric disease as defined by Diagnostic and Statistical Manual of Mental Disorders, 4th edition-Revised (DSM IV-TR, American Psychiatric Association, 2000).
5. History of surgical intervention for PD (pallidotomy, thalamotomy, deep brain stimulation, etc.).
6. Participation in a previous adenosine A2A trial.
7. Participation in any other investigational drug study within 1 month prior to randomization into this trial.
8. History of malignancy unless an exemption has been granted by the Biogen Idec Medical Director.
9. History of severe allergic or anaphylactic reactions to a drug.
10. Clinically significant cardiac, renal, pulmonary, hematopoietic, endocrine, or hepatic disease.
11. Abnormal laboratory results as follows: AST, ALT, total bilirubin, GGT levels > 1.5 x upper limit of normal; serum lipase > upper limit of normal; WBC < 4,000 cells/mm3 hemoglobin < 10, or any other abnormal laboratory value that could interfere with the assessment of safety.
12. Supine (measured in duplicate 10 minutes after resting) or standing (measured in duplicate 3 minutes after changing from a supine to a standing position) blood pressure of >150 or <90 mmHg systolic or >90 or <40 mmHg diastolic on 2 consecutive occasions.
13. Orthostatic hypotension as defined by a decrease in systolic BP of >20 mmHg or in diastolic blood pressure of > 10 mmHg measured in duplicate 3 minutes after changing from a supine to standing position.
14. History of human immunodeficiency virus (HIV).
15. Positive for hepatitis C antibody and/or positive for hepatitis B surface antigen (HBsAg) at screening.
16. History of drug or alcohol abuse as defined by the DSM IV-TR (American Psychiatric Association, 2000) within 1 year prior to randomization into this trial.
17. Alcohol use within 72 hours of Baseline Visit (Day -1).
18. Donation of blood or plasma in excess of 500 mL within 3 months of the Screening Visit.
19. Unwillingness or inability to comply with the requirements of the protocol including the presence of any condition (physical, mental, or social) that is likely to affect the subject's ability to comply with the protocol.
20. Any other reasons that, in the opinion of the Investigator and/or the Sponsor, the subject is determined to be unsuitable for enrollment in this study.

Ages: 30 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Biogen Idec, Study Director — Biogen